CLINICAL TRIAL: NCT04687644
Title: The Effect of Woman Centred Childbirth Care Training on Midwives' Patient Centred Care Competency and Job Satisfaction Levels
Brief Title: Woman Centred Childbirth Care Training
Acronym: WOCAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tuba Kızılkaya, Research assistant, Balikesir University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: A-11-21052019
Record Dates: First submitted 2020-12-27; First posted 2020-12-29 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2021-03

CONDITIONS: Childbirth Problems
Keywords: woman centred care; patient centred care competency; job satisfaction; online education

STUDY DESIGN:
Intervention Model Description: Online Education Program
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Online Education (Experimental): The education program developed within the scope of the research consists of five modules. In order to use the question and answer method in education, to make the education interactive and to receive feedback, 4 separate training groups of 7 people will be formed. The training will take place on the online platform, not face to face. Midwives will be contacted by phone and / or e-mail and the researcher will give a brief information about the research after introducing himself. A social media group will be created for each training group in order to communicate, announce trainings and inform changes.
  Interventions: Behavioral: Online education
- Control (Active Comparator): Midwives who attend the online forms of study will complete the survey. In the survey there are demographic and their view about woman centred care question forms. There are also Patient Centred Care Competency Scale and Minnesota Job Satisfaction Questionnaire. They will complete the survey.
  Interventions: Behavioral: Online education

INTERVENTIONS:
Behavioral: Online education — Education group

SUMMARY:
Woman centred childbirth care has become more meaningful and important in today's conditions. Although women-centred childbirth care is frequently mentioned in the literature, it is thought that there are no studies on this subject and it will be beneficial to train midwives on this subject. In this study, it is aimed to examine the effect of online education that will be given to midwives based on the Midwifery Model of Women-Centred Childbirth Care, on both patient-centred care competency and job satisfaction levels.

DETAILED DESCRIPTION:
Research type: Semi-experimental research -Pre-test with control group, post-test designed- Population and sample selection: The universe of the study consists of all midwives who work in the childbirth unite. The effect rate of the intervention in the research, for which the studies on the job satisfaction level of midwives are descriptive in the literature, is unknown. Therefore, Cohen standard effect rate was used. According to the sample size analysis performed in the G-Power program for the sampling, a total of 48 volunteers will be included in the study, with the power of the research being 80%, the alpha of 0.05 and the Cohen standard effect ratio of 0.8, as 26 for the intervention group and 26 for the control group. It is planned to include 52 midwives.

Hypotheses

1. Hypothesis: H0: There is no difference in patient-centered care competence levels between midwives who attended the Women-Centred Midwifery Care Training Program and those who did not.

H1: The patient-centered care competence level of midwives participating in the Women-Centred Midwifery Care Training Program is higher than the control group.

Hypothesis 2:

H0: There is no difference in job satisfaction between midwives who attended the Women-Centred Midwifery Care Training Program and those who did not.

H1: Job satisfaction of midwives participating in the Women-Centred Midwifery Care Training Program is higher than the control group.

ELIGIBILITY:
Inclusion Criteria:

* Being midwife
* Working in a childbirth unit

Exclusion Criteria:

* Midwives having a Coronavirus Disease-19 (COVID-19) infection

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-12-26 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Patient Centred Care Competency | 2 months
  Hwang et al. (2017) developed this scale. It has 4 sub-dimensions and contains 17 items. The scale is 5-point Likert type and the answers range from 1 (Strongly Disagree) to 5 (Strongly Agree).Considering the whole scale, the total Cronbach Alpha coefficient calculated as 0.850.
Job Satisfaction | 2 months
  Weiss, Davis, England ve Lofquist (1967) developed this scale. Scale is evaluated with a 5-point Likert-type scale (very satisfied- 5 points; satisfied- 4 points; indecisive- 3 points; not satisfied- 2 points; not satisfied- 1 point). In scoring, 100 is the highest score and 20 the lowest. Below 25 points indicates low job satisfaction, 26 - 74 points normal job satisfaction, 75 and above points indicate high job satisfaction. The Cronbach Alpha value was found to be 0.77.

CONTACTS AND LOCATIONS:
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No